CLINICAL TRIAL: NCT03733145
Title: A Dose Finding Trial for Angiotensin II in Hypertensive Adults on Angiotensin Converting Enzyme Inhibitors and Angiotensin Receptor Blockers With Anesthesia-Mediated Hypotension
Brief Title: Angiotensin II in General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00054661; HL-051952 (Other Grant/Funding Number: National Heart, Lung, and Blood Institute); AG070371 (Other Grant/Funding Number: National Institute on Aging)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: Angiotensin II; Angiotensin Converting Enzyme Inhibitors; Angiotensin Receptor Blockers; Anesthesia-Mediated Hypotension
MeSH Terms: conditions — Hypertension | interventions — Angiotensin II; Giapreza

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Participants on ACE inhibitors (Experimental): Participants taking ACE inhibitors (angiotensin-converting enzyme inhibitors)will be placed into this group. Intervention: Drug: Angiotensin II.
  Interventions: Drug: Angiotensin II
- Participants on ARBs (Experimental): Participants taking ARBs (angiotensin-receptor blockers) will be placed into this group. Intervention: Drug: Angiotensin II.
  Interventions: Drug: Angiotensin II
- Other Classes of Antihypertensive Agents (Experimental): Participants taking any other class of Antihypertensive Agents will be placed into this group. Intervention: Drug: Angiotensin II.
  Interventions: Drug: Angiotensin II

INTERVENTIONS:
Drug: Angiotensin II — Participants in the ACE inhibitors, angiotensin-receptor blockers (ARBs), and Other Classes of Antihypertensive Agents who's systolic blood pressure (SBP) is less than 80% of the baseline reading is detected, will have Ang II initiated at 2 ng/kg/min through a peripheral IV. The infusion will be increased at the discretion of the clinical team based on the response of the patient until a SBP within 5% of the baseline SBP.
  Other Names: Ang II; Giapreza

SUMMARY:
Hypotension in adult patients undergoing general anesthesia is common. This can lead to hypoperfusion of vital organs, organ damage, and states of increased metabolic duress. This may be worse in patients with underlying essential hypertension and worse in patients taking Angiotensin Converting Enzyme Inhibitors (ACE) and Angiotensin Receptor Blockers (ARBs). Intravenous (IV) administration of Ang II may be an effective treatment of hypotension in this patient population.

DETAILED DESCRIPTION:
Hypotension in adult patients undergoing general anesthesia is common. Many of the body's normal mechanisms to maintain adequate blood pressure in the non-anesthetized state are significantly altered by anesthetic agents, which may lead to hypotension. This can lead to hypoperfusion of vital organs, organ damage, and states of increased metabolic duress. In response to this it has become standard of care to attempt to maintain blood pressure levels within 20% of baseline in most patients under anesthesia. Maintaining the baseline blood pressure is important as patients may have pathology such as coronary artery disease, carotid stenosis, and renal artery stenosis, and hypotension may compromise the perfusion of these organs. Vasodilation also plays a key role in hypotension due to general anesthesia. Therefore, the intravenous (IV) administration of Ang II may be an effective treatment of hypotension in this patient population.The objective of this study is to determine the infusion rate of Ang II that is necessary to return systolic blood pressure (SBP) to within 5% of baseline or greater in patients with essential hypertension taking ACE inhibitors, ARBs, or different classes of antihypertensive agents and further to determine the plasma levels of different RAAS components

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension and treatment with at least one medication including an ACE inhibitor, ARB, and other agents for greater than 2 months
* Patients undergoing general anesthesia

Exclusion Criteria:

* BMI > 40
* History of deep venous thrombosis / thromboembolic disease
* History of stroke,
* Baseline SBP of ≥ 160 mmHg,
* History of myocardial infarction or cardiac stents
* Difficult airway
* Asthma
* Congestive heart failure
* Chronic obstructive pulmonary disease
* Pregnant patients

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohesh Fernando, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Comfere T, Sprung J, Kumar MM, Draper M, Wilson DP, Williams BA, Danielson DR, Liedl L, Warner DO. Angiotensin system inhibitors in a general surgical population. Anesth Analg. 2005 Mar;100(3):636-644. doi: 10.1213/01.ANE.0000146521.68059.A1. PMID 15728043
- [Background] Singh A, Antognini JF. Perioperative hypotension and myocardial ischemia: diagnostic and therapeutic approaches. Ann Card Anaesth. 2011 May-Aug;14(2):127-32. doi: 10.4103/0971-9784.81569. PMID 21636935
- [Background] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561
- [Background] Ferreira AJ, Murca TM, Fraga-Silva RA, Castro CH, Raizada MK, Santos RA. New cardiovascular and pulmonary therapeutic strategies based on the Angiotensin-converting enzyme 2/angiotensin-(1-7)/mas receptor axis. Int J Hypertens. 2012;2012:147825. doi: 10.1155/2012/147825. Epub 2012 Jan 26. PMID 22319643
- [Background] Chawla LS, Busse L, Brasha-Mitchell E, Davison D, Honiq J, Alotaibi Z, Seneff MG. Intravenous angiotensin II for the treatment of high-output shock (ATHOS trial): a pilot study. Crit Care. 2014 Oct 6;18(5):534. doi: 10.1186/s13054-014-0534-9. PMID 25286986
- [Background] Tallarida RJ, Stone DJ Jr, Raffa RB. Efficient designs for studying synergistic drug combinations. Life Sci. 1997;61(26):PL 417-25. doi: 10.1016/s0024-3205(97)01030-8. PMID 9416783

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants on ACE Inhibitors: Participants taking ACE inhibitors (angiotensin-converting enzyme inhibitors)will be placed into this group. Intervention: Drug: Angiotensin II.
  Angiotensin II: Participants in the ACE inhibitors, ARBs, and Other Classes of Antihypertensive Agents who's systolic blood pressure (SBP) is less than 80% of the baseline reading is detected, will have Ang II initiated at 2 ng/kg/min through a peripheral IV. The infusion will be increased at the discretion of the clinical team based on the response of the patient until a SBP within 5% of the baseline SBP.
- Participants on ARBs: Participants taking ARBs (angiotensin-receptor blockers) will be placed into this group. Intervention: Drug: Angiotensin II.
  Angiotensin II: Participants in the ACE inhibitors, ARBs, and Other Classes of Antihypertensive Agents who's systolic blood pressure (SBP) is less than 80% of the baseline reading is detected, will have Ang II initiated at 2 ng/kg/min through a peripheral IV. The infusion will be increased at the discretion of the clinical team based on the response of the patient until a SBP within 5% of the baseline SBP.
- Other Classes of Antihypertensive Agents: Participants taking any other class of Antihypertensive Agents will be placed into this group. Intervention: Drug: Angiotensin II.
  Angiotensin II: Participants in the ACE inhibitors, ARBs, and Other Classes of Antihypertensive Agents who's systolic blood pressure (SBP) is less than 80% of the baseline reading is detected, will have Ang II initiated at 2 ng/kg/min through a peripheral IV. The infusion will be increased at the discretion of the clinical team based on the response of the patient until a SBP within 5% of the baseline SBP.
Period: Overall Study
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Started | 10 | 11 | 11
Completed | 7 | 8 | 9
Not Completed | 3 | 3 | 2
Not completed — screenfail | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents | Total
Number analyzed (Participants) | 7 | 8 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.25 (6.16) | 67.75 (5.87) | 67.22 (6.76) | 65.29 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 4 | 4 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 9 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 6 | 6 | 7 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Dose Required to Increase the Systolic Blood Pressure (SBP)
Description: The median dose required to increase the SBP in these 3 cohorts with essential hypertension (ACE inhibitor, ARB, or those on another class of hypertensive agents) to within 5% of baseline or higher will be calculated.
Time Frame: up to 1 hour
Population: ACE Inhibitor Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol ARB Arm: 2 patients did not reach the treatment goal in this group and were therefore excluded from primary outcome analysis Other Classes of Antihypertensive Agents Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol
Measure: Median (Inter-Quartile Range); unit: ng/kg/min
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 6 | 7
ng/kg/min | 35 [35 to 45] | 43 [31 to 54] | 45 [34 to 45]

2. Secondary Outcome: Median Serum Level of Bradykinin 1-8
Description: Median serum level of Bradykinin 1-8
Time Frame: up to 1 hour
Population: ACE Inhibitor Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol Other Classes of Antihypertensive Agents Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 127043 [103938 to 180738] | 105405 [71387 to 122527] | 101169 [75851 to 130402]

3. Secondary Outcome: Median Serum Level of Bradykinin 1-7
Description: Median serum level of Bradykinin 1-7
Time Frame: Up to 1 hour
Population: ACE Inhibitor Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol Other Classes of Antihypertensive Agents: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 24457 [19026 to 35010] | 19335 [11044 to 36966] | 17438 [11906 to 25482]

4. Secondary Outcome: Median Serum Level of Bradykinin 1-5
Description: Median serum level of Bradykinin 1-5
Time Frame: Up to 1 hour
Population: ACE Inhibitor Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol Other Classes of Antihypertensive Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 2341 [1483 to 4095] | 353 [249 to 605] | 375 [251 to 534]

5. Secondary Outcome: Median Serum Level of Aldosterone
Description: Median serum level of Aldosterone
Time Frame: Up to 1 hour
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 293 [223 to 362] | 293 [223 to 362] | 230 [168 to 308]

6. Secondary Outcome: Median Serum Level of Angiotensin I
Description: Median serum level of Angiotensin I
Time Frame: Up to 1 hour
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 8.7 [0 to 37.9] | 1.8 [0 to 16.7] | 0 [0 to 6.3]

7. Secondary Outcome: Median Serum Level of Angiotensin II
Description: Median serum level of Angiotensin II
Time Frame: up to 1 hour
Population: ACE Inhibitors Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol Other Classes of Antihypertensive Agents Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 10.9 [3.7 to 370.1] | 31.2 [5 to 758.5] | 10.2 [0 to 326.2]

8. Secondary Outcome: Median Serum Level of Angiotensin IV
Description: Median serum level of Angiotensin IV
Time Frame: Up to 1 hour
Population: ACE Inhibitors Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol Other Classes of Antihypertensive Agents: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 0 [0 to 11] | 1 [0 to 18.7] | 0 [0 to 8.2]

9. Secondary Outcome: Median Serum Level of Angiotensin 1-7
Description: Median serum level of Angiotensin 1-7
Time Frame: Up to 1 hour
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 8.7 [0 to 37.9] | 1.8 [0 to 16.7] | 0 [0 to 6.3]

10. Secondary Outcome: Median Serum Level of Angiotensin 1-5
Description: Median serum level of Angiotensin 1-5
Time Frame: Up to 1 hour
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 0 [0 to 0] | 0 [0 to 28.8] | 0 [0 to 0]

11. Secondary Outcome: Median Serum Level of Angiotensin 1-9
Description: Median serum level of Angiotensin 1-9
Time Frame: Up to 1 hour
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

12. Secondary Outcome: Median Serum Level of Angiotensin 2-10
Description: Median serum level of Angiotensin 2-10
Time Frame: Up to 1 hour
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 0 [0 to 5.8] | 0 [0 to 0] | 0 [0 to 0]

13. Secondary Outcome: Median Serum Level of Angiotensin 2-7
Description: Median serum level of Angiotensin 2-7
Time Frame: Up to 1 hour
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

14. Secondary Outcome: Median Serum Level of Angiotensin 3-7
Description: Median serum level of Angiotensin 3-7
Time Frame: Up to 1 hour
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 5 | 8 | 7
pmol/L | 0 [0 to 2.33] | 0 [0 to 0] | 0 [0 to 0]

15. Secondary Outcome: Median Serum Level of Angiotensin 1-12
Description: Median serum level of Angiotensin 1-12
Time Frame: Up to 1 hour
Population: ACE Inhibitors Arm: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol, 2 patients unable to get sample.
  ARBs Arm: 1 patient unable to get sample. Other Classes of Antihypertensive Agents: 2 patients did not experience hypotension and therefore did not receive the Ang II per protocol, 2 patients unable to get sample.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
Number analyzed (Participants) | 3 | 7 | 5
pmol/L | 940 [788 to 982] | 1011 [846 to 1138] | 674 [344 to 1043]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Participants on ACE Inhibitors | Participants on ARBs | Other Classes of Antihypertensive Agents
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/5 | 2/8 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants on ACE Inhibitors (N=5) | Participants on ARBs (N=8) | Other Classes of Antihypertensive Agents (N=7)
Leg Swelling (Vascular disorders) | 1 | 0 | 0
Blurred Vision (Eye disorders) | 0 | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — arthritic shoulder and arm pain from surgery positioning
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT03733145/Prot_SAP_002.pdf
  • Informed Consent Form (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT03733145/ICF_001.pdf